CLINICAL TRIAL: NCT03581292
Title: A Phase 2 Study of Veliparib (ABT-888) and Local Irradiation, Followed by Maintenance Veliparib and Temozolomide, in Patients With Newly Diagnosed High-Grade Glioma (HGG) Without H3 K27M or BRAFV600 Mutations
Brief Title: Veliparib, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed Malignant Glioma Without H3 K27M or BRAFV600 Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01361; NCI-2018-01361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1721 (Other: Children's Oncology Group); ACNS1721 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2018-07-04; First posted 2018-07-10 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-07

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma; Malignant Glioma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Radiotherapy; Radiation; Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, veliparib, temozolomide) (Experimental): CHEMORADIOTHERAPY PHASE: Patients receive veliparib PO BID and undergo 30 daily fractions of radiation therapy 5 days per week for 6-7 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE CHEMOTHERAPY: Beginning 4 weeks after chemoradiotherapy phase, patients receive veliparib PO BID and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide; Drug: Veliparib

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase II trial studies how well veliparib, radiation therapy, and temozolomide work in treating patients with newly diagnosed malignant glioma without H3 K27M or BRAFV600 mutations. Poly adenosine diphosphate (ADP) ribose polymerases (PARPs) are proteins that help repair DNA mutations. PARP inhibitors, such as veliparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib, radiation therapy, and temozolomide may work better in treating patients with newly diagnosed malignant glioma without H3 K27M or BRAFV600 mutations compared to radiation therapy and temozolomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether veliparib (ABT-888), when added to radiotherapy (RT) and temozolomide, is efficacious for the treatment of patients with newly-diagnosed high-grade glioma (HGG) whose tumors' molecular profile are wild-type for H3 K27M, BRAF, and IDH1/2.

II. To determine whether veliparib (ABT-888), when added to RT and temozolomide, is efficacious for the treatment of patients with newly-diagnosed HGG whose tumors' molecular profile are wild-type for H3 K27M and BRAF and harbor an IDH1/2 mutation.

EXPLORATORY OBJECTIVES:

I. To explore associations of genomic, transcriptomic, and/or epigenetic alterations of the tumors with treatment response and outcome.

II. To explore the extent to which patients with BRCA1/2 gene alterations and other deoxyribonucleic acid (DNA) damaged genes display tumor genomic features consistent with homologous repair deficiency (HRD), including large scale state transitions (LSTs), mutational signature 3, and an enrichment for deletions flanked by sequences of (micro) homology.

III. To explore the burden of high, moderate, and low penetrant germline alterations in HRD genes (such as BRCA1, BRCA2, PALB2, Fanconi complex genes, ATM, CHEK2, RAD51B/C/D), mis-match repair genes (such as MLH1, MSH2, MSH6, PMS2, EPCAM), and energy metabolism genes (such as SDHA, SDHB, SDHC, SDHAF2, SDHD, IDH1, IDH2, and FH).

IV. To explore constitutional imprinting abnormalities associated with EP300 and IGF2 in peripheral blood from patients with HGGs.

OUTLINE:

CHEMORADIOTHERAPY PHASE: Patients receive veliparib orally (PO) twice daily (BID) and undergo 30 daily fractions of radiation therapy 5 days per week for 6-7 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CHEMOTHERAPY: Beginning 4 weeks after chemoradiotherapy phase, patients receive veliparib PO BID and temozolomide PO once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for year 1, every 4 months for year 2, every 6 months for year 3, and then once yearly for years 4-10.

ELIGIBILITY:
Inclusion Criteria:

* Stratum 1 (IDH wild-type): Patients must be >= 3 years of age and =< 21 years of age at the time of enrollment

  * Please note Stratum 1 was closed to accrual on January 24, 2020
* Stratum 2 (IDH mutant): Patients must be >= 3 years of age and =< 25 years of age at the time of enrollment
* Patients must have eligibility confirmed by rapid central pathology and central molecular screening reviews performed on APEC14B1:

  * Newly-diagnosed high-grade glioma such as anaplastic astrocytoma or glioblastoma
  * Negative results for H3 K27M by immunohistochemistry (IHC)
  * Negative results for BRAFV600 mutation by next-generation sequencing (NGS)
* Patients must have histological verification of diagnosis. Patients with M+ disease (defined as evidence of neuraxis dissemination) are not eligible. Cerebrospinal fluid (CSF) cytology is not required but may be obtained if clinically indicated prior to study enrollment. If cytology is positive, the patient would be considered to have metastatic disease and would, therefore, be ineligible
* Pre-operative and post-operative brain magnetic resonance imaging (MRI) with and without contrast must be obtained. The requirement for a post-operative MRI is waived for patients who undergo biopsy only. A spine MRI is not required, but may be obtained if clinically indicated. If the spine MRI is positive, the patient would be considered to have M+ disease (defined as neuraxis dissemination) and would be ineligible
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Peripheral absolute neutrophil count (ANC) >= 1,000/uL (within 7 days prior to enrollment)
* Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to enrollment)
* Hemoglobin >= 8.0 gm/dL (can be transfused) (within 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * 3 to < 6 years: 0.8 (male and female) maximum serum creatinine (mg/dL)
  * 6 to < 10 years: 1 (male and female) maximum serum creatinine (mg/dL)
  * 10 to < 13 years: 1.2 (male and female) maximum serum creatinine (mg/dL)
  * 13 to < 16 years: 1.5 (male), 1.4 (female) maximum serum creatinine (mg/dL)
  * >= 16 years: 1.7 (male), 1.4 (female) maximum serum creatinine (mg/dL)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L
* Patients with seizure disorder may be enrolled if seizures are well-controlled (i.e., patients must not have required rescue medications for uncontrolled seizures within 14 days prior to enrollment)
* Patients must be enrolled and protocol therapy must be projected to begin no later than 31 days after definitive surgery (Day 0). If a biopsy only was performed, the biopsy date will be considered the date of definitive surgery. For patients who have a biopsy or incomplete resection at diagnosis followed by additional surgery, the date of the last resection will be considered the date of definitive surgery
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with the following histologies:

  * Diffuse astrocytoma (grade 2)
  * Oligodendrogliomas (any grade)
  * Pleomorphic xanthoastrocytoma (PXA, any grade)
* Patients with primary tumor location of brainstem or spinal cord
* Patients with M+ disease (defined as neuraxis dissemination either by imaging or by cytology)
* Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/myelodysplastic syndrome (MDS) or with features suggestive of AML/MDS
* Prior allogenic bone marrow transplant or double umbilical cord blood transplantation
* Patients must not have received any prior tumor-directed therapy including radiation therapy, chemotherapy (tumor-directed therapy), molecularly targeted agents, or immunotherapy for the treatment of HGG other than surgical intervention and/or corticosteroids
* Lumbar CSF cytology is not required, but may be performed if clinically indicated prior to study enrollment. If lumbar CSF cytology is positive, the patient is considered to have M+ disease and is ineligible

  * Note: False positive cytology can occur within 10 days of surgery
* Patients with gliomatosis cerebri type 1 or 2
* Patients who are not able to receive protocol specified radiation therapy
* Patients must not be currently receiving other anti-cancer agents
* Patients with known constitutional mismatch repair deficiency syndrome (CMMR-D)/biallelic mismatch repair deficiency (bMMRD)
* Female patients who are pregnant are ineligible due to risks of fetal and teratogenic adverse events as seen in animal/human studies
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for 6 months after the last dose of protocol-specified chemotherapy

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-10-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Karajannis, Principal Investigator — Children's Oncology Group
Locations (163):
- United States (145):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

REFERENCES:
- [Derived] Karajannis MA, Onar-Thomas A, Lin T, Baxter PA, Boue DR, Cole BL, Fuller C, Haque S, Jabado N, Lucas JT Jr, MacDonald SM, Matsushima C, Patel N, Pierson CR, Souweidane MM, Thomas DL, Walsh MF, Zaky W, Leary SES, Gajjar A, Fouladi M, Cohen KJ. Phase 2 trial of veliparib, local irradiation, and temozolomide in patients with newly diagnosed high-grade glioma: a Children's Oncology Group study. Neuro Oncol. 2025 May 15;27(4):1092-1101. doi: 10.1093/neuonc/noae247. PMID 39560182

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1: Pediatric newly-diagnosed HGG patients who are wild-type with respect to H3 K27M, BRAF, and IDH1/2
- Stratum 2: Pediatric newly-diagnosed HGG patients who are positive for either IDH1/2 mutation
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 24 | 14
Completed | 11 | 9
Not Completed | 13 | 5
Not completed — Physician Decision | 9 | 5
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Withdrawal before Therapy Start | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 24 | 14 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 6 | 29
  Between 18 and 65 years | 1 | 8 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (4) | 18.4 (2.9) | 14.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 20 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 12 | 31
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 13 | 29
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: Compare event free survival to historical data for each stratum. Analysis will be based on a 2-sample, 1 sided logrank test. EFS is measured from time of enrollment to the date of first documented progression, second malignancy, or date of death from any cause, whichever comes first. Subjects who do not have any event will be censored at the last follow-up date.
Time Frame: Up to 2 years
Population: Participants who received study therapy will be included in the analysis.
Measure: Number; unit: probability
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 23 | 14
probability | 0.9857 | 0.9571

2. Secondary Outcome: Objective Response
Description: Estimate the objective response rate in patients with measurable disease. The 95% confidence interval will be calculated by Clopper-Pearson method. Objective responses are defined as patients who achieved complete response or partial response anytime during treatment. Tumor response criteria are determined by changes in size using the longest tumor dimension, and its perpendicular. Either T1, T2 weighted/FLAIR images are used - whichever gives the best estimate of tumor size. Complete Response (CR): Disappearance of all target lesions; Partial response (PR): >=50% decrease in the sum of the products of the two perpendicular diameters of target lesions, compared to baseline measurement. Objective Response = CR + PR.
Time Frame: Anytime during treatment (up to 1 year from enrollment)
Population: Participants who had measurable disease at baseline and received study therapy will be included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 11 | 7
percentage of participants | 9.1 [0.2 to 41.3] | 14.3 [0.4 to 57.9]

3. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate the 2-year overall survival for each stratum. OS is measured from time of enrollment to the date of death from any cause. Subjects who do not have any event will be censored at the last follow-up date.
Time Frame: Up to 2 years
Population: Participants who received study therapy will be included in the analysis.
Measure: Number (95% Confidence Interval); unit: survival probability of patients
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 23 | 14
survival probability of patients | 0.27 [0.11 to 0.46] | 0.85 [0.52 to 0.96]

4. Other Pre Specified Outcome: Biomarker Analysis
Description: Will provide a frequency table summarizing the number of patients with each aberration/alteration detected in germline and/or tumor samples. For longitudinal plasma samples used to assess circulating tumor deoxyribonucleic acid, will summarize the percentage of patients with samples as well as display/summarize any changes in molecular markers. When feasible we will explore the association of these aberrations with EFS/OS and objective response rates via Cox models and fisher exact tests, respectively. Will also explore associations between genetic variants and clinical/demographic variables including age, resection status, histology, etc. For analyses exploring associations of a large number of potential markers with clinical outcome, will utilize false discovery rate approaches in order to control family-wise error rate.
Time Frame: Up to 5.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment up to 3 years after enrollment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Stratum 1 | Stratum 2
All-Cause Mortality (participants affected / at risk) | 18/23 | 3/14
Serious Adverse Events (participants affected / at risk) | 22/23 | 5/14
Other Adverse Events (participants affected / at risk) | 4/23 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=23) | Stratum 2 (N=14)
Death NOS (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 16 (16) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (7) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 4 (4) | 2 (3)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
entrapped ventricle (Nervous system disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=23) | Stratum 2 (N=14)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03581292/Prot_SAP_000.pdf